CLINICAL TRIAL: NCT05262556
Title: Pilot Study of NP-101 (TQ Formula) in Combination With Nivolumab and Ipilimumab in Advanced and Metastatic Extra-pulmonary Neuroendocrine Carcinomas (EP-NECAs)
Brief Title: NP-101 (TQ Formula) With Nivolumab and Ipilimumab in Advanced or Metastatic Extra-pulmonary Neuroendocrine Carcinomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amr Mohamed MD (Other)
Collaborators: Novatek Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Amr Mohamed MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5221
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor; Gastroenteropancreatic Neuroendocrine Neoplasm; Neuroendocrine Carcinoma; Mixed Neuroendocrine-Non Neuroendocrine Neoplasm
Keywords: Extrapulmonary Neuroendocrine Carcinoma
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Carcinoma, Neuroendocrine | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NP-101 (TQ Formula) + Nivolumab + Ipilimumab (Experimental)
  Interventions: Drug: NP-101 (TQ Formula); Drug: Nivolumab (3mg/kg); Drug: Ipilimumab (1mg/kg)

INTERVENTIONS:
Drug: NP-101 (TQ Formula) — Oral, five 600mg tabs daily every three weeks for four cycles (21-day cycle), then maintenance for an additional 12 weeks for a total of six cycles.
  Other Names: Black seed oil capsules
Drug: Nivolumab (3mg/kg) — Intravenously on Day 1 every three weeks for four cycles (maximum dose 360mg once every 3 weeks), then 240mg maintenance every two weeks for six cycles for a total of six months of treatment.
  Other Names: Opdivo
Drug: Ipilimumab (1mg/kg) — Intravenously on day 1 of each (21-day) cycle for a total of four cycles only.
  Other Names: Yervoy

SUMMARY:
A pilot study to evaluate the anti-tumor efficacy of this novel combined regimen (NP-101 TQ Formula plus nivolumab and ipilimumab) in the second-line setting for EP-NECA. NP-101 (TQ Formula) (TQ, C10H12O2) is the main bioactive component of the black seed (Nigella sativa, Ranunculaceae family) and has anti-oxidant, anti-angiogenic effects.

DETAILED DESCRIPTION:
The purpose of this study is to find out if NP-101 (TQ Formula) given with the immunotherapy drugs called nivolumab and ipilimumab helps with neuroendocrine carcinoma who have progressed on at least one first line standard therapy. NP-101 (TQ Formula) black seed oil tablet is an investigational (experimental) drug that may enhance the effect that immunotherapy drugs such as nivolumab and ipilimumab have on neuroendocrine carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed of relapsed and/or refractory unresectable advanced and/or metastatic high-grade extra-pulmonary neuroendocrine carcinoma (EP-NECAs), and have failed at least one standard line of therapy.
* Subjects must have received at least one prior therapy for this disease. Subjects must have recovered from acute toxicities of prior chemotherapy. Any prior non-hematologic vital organ toxicity (cardiac, pulmonary, hepatic, and renal) of previous therapy must have resolved to grade 1 or less. Neurological toxicities must have resolved to grade 2 or less.
* Age >18 years.
* Subjects must have radiologic disease measurable by RECIST criteria.
* All previous chemotherapy or radiation must be completed at least three weeks prior to starting study treatment.
* Performance status ECOG Performance status ≤ 2
* Subjects must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 7.0 g/dl
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 75,000/mcL
  * Total bilirubin ≤ 3 X institutional upper limit of normal (except subjects with elevated bilirubin unrelated to liver dysfunction)
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine ≤ 1.5 X institutional upper limit of normal
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Subjects of childbearing potential must agree to practice reliable contraception or to practice abstinence for at least 28 days before and for 60 days after the last dose of study drug. Reliable contraception is defined as:

  * One highly effective method and one additional effective (barrier) method:
  * Examples of highly effective methods:
* Intrauterine device (IUD)
* Hormonal (injections, implants, levonorgestrel-releasing intrauterine system [IUS], medroxyprogesterone acetate depot injections, ovulation inhibitory progesterone-only pills [e.g. desogestrel])
* Tubal ligation
* Partner's vasectomy

  * Examples of additional effective methods:
* Male condom
* Diaphragm
* Cervical Cap

Inclusion of Women and minorities

* People of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Well-differentiated GEP-NETs are excluded from this trial.
* Prior treatment toxicities that have not resolved to ≤ Grade 2 according to NCI CTCAE Version 5.0 (list exceptions, e.g. alopecia, neuropathy, etc).
* Subjects received prior nivolumab or ipilimumab
* Subjects with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with treated oligometastatic CNS metastases will be considered for the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to NP-101 (TQ Formula) or immunotherapy (nivolumab or ipilimumab) used in this study.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because NP-101 (TQ Formula) effects on pregnancy and the fetus used in this protocol is unknown.
* Known chronic active untreated hepatitis B or C infection.
* HIV-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with NP-101 (TQ Formula) and immunotherapy agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Antitumor activity of NP-101 (TQ Formula) plus nivolumab and ipilimumab in subjects with advanced and/or metastatic EP-NECAs who progressed on first line therapy | Up to 6 months from the start of treatment
  Antitumor activity will be measured by the number of participants that have a complete response (CR), partial response (PR), or stable disease (SD). CR is defined as the complete disappearance of all target lesions, confirmed by repeat assessments at no less than 4 weeks after the criteria for response is first met. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum longest diameter. SD is defined as neither sufficient decrease to qualify for a partial response nor sufficient increase to qualify for progressive disease.

SECONDARY OUTCOMES:
Safety profile/toxicity of combining NP-101 (TQ Formula) with nivolumab and ipilimumab. | Up to 2 years from the start of treatment
  Number of participants who experience a Grade 3 or greater drug-related adverse events.
Time to progression (TTP) | Up to 6 months from the start of treatment
  To determine the time to progression (TTP) using NP-101 (TQ Formula) plus nivolumab and ipilimumab combined regimen in subjects with EP-NECAs

CONTACTS AND LOCATIONS:
Overall Officials: Amr Mohamed, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States